CLINICAL TRIAL: NCT02097459
Title: Prognostic Evaluation of Changing Endocrine Therapy in Perimenopausal and Recently Postmenopausal Women With Early-stage Hormone Receptor-Positive Breast Cancer
Brief Title: Prognostic Evaluation of Changing Endocrine Therapy in Women With Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Qiang SUN, Chief of Breast Surgery Department, Professor, Peking Union Medical College Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PUMCH-BREAST-AI
Record Dates: First submitted 2014-03-19; First posted 2014-03-27 (Estimated); Last update posted 2016-05-25 (Estimated); Status verified 2016-05

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Endocrine therapy; Perimenopausal and recently postmenopausal patients; Early-stage hormone receptor-positive
MeSH Terms: conditions — Breast Neoplasms | interventions — Anastrozole; Tamoxifen; Toremifene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Failed group (Experimental): Patients who have recurrence of menstruation after changing endocrine therapy to anastrozole and then go back to the original SERMs therapy.
  Interventions: Drug: Anastrozole; Drug: Tamoxifen; Drug: Toremifene
- Succeeded group (Experimental): Patients who have no recurrence of menstruation after changing endocrine therapy and then go on with anastrozole therapy.
  Interventions: Drug: Anastrozole
- No chang group (Active Comparator): Patients who don't change the endocrine therapy and go on with the original tamoxifen or toremifene therapy.
  Interventions: Drug: Tamoxifen; Drug: Toremifene

INTERVENTIONS:
Drug: Anastrozole
  Other Names: Arimidex
  Arms: Failed group; Succeeded group
Drug: Tamoxifen
  Arms: Failed group; No chang group
Drug: Toremifene
  Other Names: Fareston; Shu Rui
  Arms: Failed group; No chang group

SUMMARY:
It suggests in the Guideline that the postmenopausal women with breast cancer who have taken selective estrogen receptor modulators (SERMs) therapy for 2-3 years could benefit from changing endocrine therapy to aromatase inhibitors (AIs). This is a prospective, randomized and non-inferior trial to evaluate the prognosis of changing endocrine therapy from SERMs to AIs in perimenopausal and recently postmenopausal women with early-stage hormone receptor-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent must be obtained and documented according to the local regulatory requirements prior to beginning specific protocol procedures.
* Age of at least 45 and at most 55 years.
* Performance status (Karnofsky-Index) >80%
* Steroid receptor (estrogen and progesterone) positive tumor (diagnosis according to hospital standard-procedures).
* No clinical evidence of local recurrence or distant metastases.
* Complete staging work-up within 3 months prior to registration. All patients must have (bilateral) mammography or breast MRI, chest X-ray; other tests may be performed as clinically indicated.
* Patients have taken the SERMs as endocrine therapy for 2-4 years.
* Patients who have had amenorrhea for at least half a year.
* Life expectancy of at least 10 years, disregarding the diagnosis of cancer.
* Adequate organ function including normal red and white blood count, platelets, serum creatinine, bilirubin, and transaminases within normal range of the institution.
* Patients must be available for and compliant to treatment and follow-up.
* Patients registered on this trial must be treated and followed up at the participating center.

Exclusion Criteria:

* Known hypersensitivity reaction to the investigational compounds or incorporated substances.
* Hormone receptor-negative breast cancer.
* Local recurrence and/or metastasis of breast cancer.
* History of hysterectomy.
* Pregnant or lactating patients. Patients of childbearing potential must have a negative pregnancy test (urine or serum) within 14 days prior to registration.
* History of osteoporosis and/or fractures due to osteoporosis.
* Prior or concomitant secondary malignancy (except non-melanomatous skin cancer or carcinoma in situ of the uterine cervix)
* Any other serious medical pathology, such as congestive heart failure; unstable angina; history of myocardial infarction during the previous year; uncontrolled high risk arrhythmias
* Other serious illness or medical condition that may interfere with the understanding and giving of informed consent and the conduct of the study.
* Concurrent treatment with other experimental drugs or any other anti-cancer therapy.
* Males.

Ages: 45 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Estimated)
Dates: Start 2014-03; Primary Completion 2024-03 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | 10 years
Overall Survival | 10 years

SECONDARY OUTCOMES:
Disease Free Survival | 5 years
Overall Survival | 5 years

OTHER OUTCOMES:
Disease Free Survival | 3 years
Overall Survival | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Sun, Doctor, Study Chair — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, China